CLINICAL TRIAL: NCT02465125
Title: The Transfusion Triggers in Vascular Surgery Trial: Two Different Transfusion Triggers for Postoperative Haemoglobin Separation and Adherence to Transfusion Strategies in Vascular Surgery: a Randomised Clinical Feasibility Trial
Brief Title: The Transfusion Triggers in Vascular Surgery Trial
Acronym: TV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Naestved Hospital (Other)
Collaborators: Copenhagen Trial Unit, Center for Clinical Intervention Research (Other); Research Unit, Naestved, Region Zealand, Denmark. (Unknown)
Responsible Party: Principal Investigator, Anders Møller, Resident, Slagelse Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SJ-426
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Atherosclerosis; Anemia; Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases
MeSH Terms: conditions — Atherosclerosis; Anemia; Aortic Aneurysm, Abdominal; Arterial Occlusive Diseases | interventions — Erythrocyte Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low transfusion trigger (Active Comparator): Intervention group. Low or restrictive transfusion trigger: hemoglobin < 5 mmol/L (approx. 8 g/dl or a hematocrit of 25%) This trigger is what is recommended by the Danish Health and Medicines Authority for stable patients with chronic heart disease.
  Interventions: Biological: red blood cell transfusion
- High transfusion trigger (Active Comparator): Control group. High or liberal transfusion trigger: hemoglobin < 6 mmol/L (approx. 10 g/dl or a hematocrit of 30%) This trigger reflects the practice among Danish vascular anesthesiologists and correspond to the transfusion trigger recommended by the European society for vascular surgery
  Interventions: Biological: red blood cell transfusion

INTERVENTIONS:
Biological: red blood cell transfusion
  Other Names: erythrocyte transfusion

SUMMARY:
BACKGROUND

* Vascular surgical patients often receive red blood cell (RBC) transfusions in the peri-operative period
* RBC transfusion may lead to improved outcome but on the other hand the intervention may be harmful
* Danish Health and Medicines Authority recommends transfusion of RBC at hemoglobin below 5 mmol/L while local clinical guidelines recommend transfusion of RBC to maintain hemoglobin levels above 6 mmol/L
* A large randomized clinical trial is needed to evaluate the efficacy and safety of RBC transfusion in patients undergoing vascular surgery.
* A trial examining the effect of RBC transfusion on tissue oxygenation is used to test the trial-design and feasibility for a trial evaluating post-operative mortality and morbidity.

DETAILED DESCRIPTION:
DESIGN Single-center, randomized, open-label trial including vascular surgical patients for peri-operative red blood cell (RBC) transfusion.

If the patient drops out of the trial, either at his/her own request or due to withdrawal from active therapy, the patient will be followed up in the intention-to-treat analyses.

PROTOCOL SUSPENSION

The patient can temporarily be suspended from the protocol in the following circumstances, if the clinician in charge finds indication for blood transfusions not adhering to the planned transfusion threshold:

* Uncontrollable bleeding, defined as loss of surgical hemostasis resulting in overt or imminent hemodynamic instability with insufficient tissue oxygenation and increasing lactate production OR
* Hypotension unresponsive to fluid replacement OR
* Decompensated heart failure OR
* Stroke, extremity- and intestinal ischaemia

SAMPLE SIZE With a total of 50 randomised patients, the trial is powered to

* Show difference in mean postoperative hemoglobin of 1.0 mmol/L. With a power of 95%, 5% significance and a standard deviation of 0.9 mmol/L.
* Show a difference in 2 units (600 mL) of RBC transfused based on a standard deviation of RBC transfusion volume of 717 mL, with a power of 80 % and 5% significance
* Produce a 97.5% confidence interval (CI) equal to the sample adherence prevalence plus or minus 8% when the true prevalence of adherence is hypothesized to be 90%
* Detect a difference in near infrared spectroscopy-determined tissue oxygenation (ScO2) of 6 % during surgery. With a power of 80%, 5% significance and a ScO2-standard deviation of 7%

TIME-LINE The first patient is expected to be randomized June 8th 2015, the last will be randomized March 31st 2016 and the trial database is expected to be closed ultimo June 2016. The main manuscript will be submitted shortly thereafter.

PROTOCOL AMENDMENTS

1. The Ethical Committee of Region Zealand has approved a protocol amendment of March 29th 2016 for permission of extending the trial period to the end of 2016.
2. On September 20th 2016 The Ethical Committee of Region Zealand approved a protocol amendment of September 16th 2016 for permission of extending the sample size to 58 patients and extending the trial period to June 31st 2017.

The 2nd amendment was submitted to compensate for an unexpected high rate of patients randomised postoperatively and thus to secure a sufficient sample size (n=44) for the primary outcome measure, postoperative Hb, and the secondary outcome measures NIRS and ROTEM.

ELIGIBILITY:
Inclusion Criteria:

* Patients for planned open repair of the abdominal aorta or infrainguinal arterial bypass
* Hemoglobin < 6 mmol/L

Exclusion Criteria:

* Documented wish against transfusion
* Previous serious adverse reaction with blood products
* Unable to understand the benefits and risks of testing
* Previous participation in trial

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-07-15 (Actual); Primary Completion 2016-12-08 (Actual); Study Completion 2017-01-09 (Actual)

PRIMARY OUTCOMES:
Mean Post-operative hemoglobin (longitudinal outcome) | Day 0 - 15
  Day 0 is the hemoglobin measured upon arrival at the recovery room or at the intensive care unit depending on what level of care the patient needs after surgery.

SECONDARY OUTCOMES:
Units of red blood cells transfused (count data) | 30 days after operation
  During 30 day trial period
Recruitment rate with 95% confidence interval | Day -1 (day before operation)
  Defined as the ratio of: number of patients included divided by the number of patients eligible (fulfilling the inclusion criteria)
Protocol suspension | 30 days after operation
  Number of patients having their protocol suspended after primary inclusion due to hemodynamic instability
Protocol adherence | 30 days after operation
  Adherence to hemoglobin concentrations used for transfusion triggers
Intraoperative tissue oxygenation | Participants will be monitored during their stay at the operation theatre, an expected average of 3 hours
  The outcome measure is defined as lowest values and area-under-baseline calculations. Baseline is defined as the average saturation value over a 1-min period after the patient has been fluid optimized after induction of anesthesia, before start of surgery.
Changes in coagulation competence measured by rotational thromboelastometry (ROTEM) | An expected average time frame of 3 hours
  Changes in coagulation competence will be the baseline ROTEM level (before induction of anesthesia) compared to the end of surgery ROTEM level.
Severe adverse events | 30 days after operation
  myocardial injury, acute kidney injury, 30-days mortality, ischemic stroke, severe adverse transfusion reactions
Explorative Outcomes | 90 days after operation
  1. Major cardiovascular events (acute myocardial infarction, stroke, renal replacement therapy, vascular reoperation and amputation) (dichotomous outcome) AND
  2. Days alive outside hospital within 90 days (count data)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Møller, Resident, Principal Investigator — Slagelse Hospital
Locations (1):
- Slagelse Hospital, Slagelse, Region Sjælland, Denmark

REFERENCES:
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Fergusson DA, Pagano MB, Roubinian NH, Turgeon AF, Valentine S, Trivella M, Doree C, Hebert PC. Transfusion thresholds and other strategies for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2025 Oct 20;10(10):CD002042. doi: 10.1002/14651858.CD002042.pub6. PMID 41114449
- [Derived] Carson JL, Stanworth SJ, Dennis JA, Trivella M, Roubinian N, Fergusson DA, Triulzi D, Doree C, Hebert PC. Transfusion thresholds for guiding red blood cell transfusion. Cochrane Database Syst Rev. 2021 Dec 21;12(12):CD002042. doi: 10.1002/14651858.CD002042.pub5. PMID 34932836
- [Derived] Moller A, Nielsen HB, Wetterslev J, Pedersen OB, Hellemann D, Winkel P, Marcussen KV, Ramsing BGU, Mortensen A, Jakobsen JC, Shahidi S. Low vs high hemoglobin trigger for transfusion in vascular surgery: a randomized clinical feasibility trial. Blood. 2019 Jun 20;133(25):2639-2650. doi: 10.1182/blood-2018-10-877530. Epub 2019 Mar 11. PMID 30858230